CLINICAL TRIAL: NCT07365579
Title: mHealth for Suicide Prevention: Design, Development, and Feasibility of a Scalable SMS-based Safety Planning Intervention
Brief Title: Design and Feasibility of an SMS-based Safety Planning Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jonah Meyerhoff, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STU00217191; K08MH128640 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation and Behavior
Keywords: Text message; safety plan; suicide prevention
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: enhanced waitlist control design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS based safety planning intervention (SMS-SPI) (Experimental): The SMS-SPI consists of a 4-week automated text messaging intervention. It is designed to guide users through the steps of the safety planning process for management of suicide related thoughts and behaviors. The intervention delivers structured, interactive messages daily addressing coping strategies, crisis resources, environmental safety, family and friends for support, distraction techniques, and recognition of warning signs. The number of messages sent each day varies based on users' interactions with the program; users who respond more frequently may receive more messages. In addition to text messaging, the program includes a web-based interface that enabled users to conveniently review and update their safety plan. The SMS-SPI uses message stems that establish a particular topic (e.g., identification of crisis warning signs) and message probes that follow-up on users' responses, which is individualized through branching logic.
  Interventions: Behavioral: Text Messaging based Safety Planning Intervention
- Enhanced waitlist control (eWLC) (Active Comparator): Text messages that are non-interactive and contain referral to crisis services (e.g., the National Suicide Prevention Lifeline, the Crisis Text Line, and (c) the Trevor Project Lifeline). Facilitated referral is a first-line prevention strategy for suicide and is a best-practice commonly integrated into internet-based screenings and informational tools.
  Interventions: Behavioral: Text Messaging based Safety Planning Intervention; Behavioral: Facilitated Referral to Crisis Resources

INTERVENTIONS:
Behavioral: Text Messaging based Safety Planning Intervention — A 4-week automated text messaging intervention designed to guide users through the steps of the safety planning process. The intervention delivers structured, interactive messages daily addressing coping strategies, crisis resources, environmental safety, family and friends for support, distraction techniques, and recognition of warning signs.
Behavioral: Facilitated Referral to Crisis Resources — Text messages that are non-interactive and contain referral to crisis services (e.g., the National Suicide Prevention Lifeline, the Crisis Text Line, and (c) the Trevor Project Lifeline).
  Arms: Enhanced waitlist control (eWLC)

SUMMARY:
This study is testing whether it is feasible to run a larger randomized controlled trial and whether an automated text messaging program is acceptable to young adults who have suicidal thoughts. The program is designed to help participants create and use a safety plan, which is a personalized list of warning signs, coping strategies, supportive people, professional resources, ways to make their environment safer, and reasons for living. After joining and completing an initial survey, participants are randomly assigned by a computer to one of two groups. One group starts right away with the interactive safety planning text program. The other group first receives simple text messages with 24/7 crisis resources and then, after four weeks, also receives the interactive safety planning program. Participants use the text program for about four weeks and complete online surveys at the start and again over a total period of 24 weeks.

DETAILED DESCRIPTION:
This study is a randomized, controlled feasibility trial testing an automated text messaging program designed to help young adults (ages 18 to 24) who have recently experienced suicidal thoughts create and use a personalized safety plan. A safety plan is a step-by-step list of warning signs, coping strategies, supportive people, professional resources, ways to make the environment safer, and personal reasons for living that can be used during times of crisis. The main goals of the study are not to prove effectiveness or efficacy, but to determine whether it is possible to run a larger randomized controlled trial in the future and whether young adults find this type of text-based safety planning acceptable, usable, and engaging.

Sixty participants will be enrolled from across the United States through Mental Health America and online outreach. After completing screening, providing consent, finishing baseline surveys, and confirming they can receive text messages, participants will be randomly assigned by a computer, like flipping a coin, to one of two groups. Neither participants nor study staff choose the group assignment. One group will receive the interactive safety-planning text program right away. The other group will first receive supportive but non-interactive text messages that provide 24/7 crisis resources, and after four weeks will also begin the same interactive safety-planning program. This "enhanced waitlist" design allows all participants to eventually receive the intervention while still allowing researchers to compare early outcomes between groups.

The interactive program lasts four weeks and sends daily text messages that guide users through building and practicing their safety plan. Messages ask participants to reflect on their own experiences, write responses in their own words, identify coping activities, supportive people, crisis services, and ways to reduce access to dangerous means. The system uses follow-up questions and branching logic so that each person's safety plan becomes detailed and highly personalized. Participants can also review and update their plan through a secure web link and can request different modules on demand. After the four-week active phase, participants can continue to access their safety plan for the rest of the 24-week study period.

Throughout the study, participants complete online surveys at the start and again at 2, 4, 8, 16, and 24 weeks. These surveys measure suicidal thoughts and behaviors, coping skills, emotional pain, hopelessness, social connection, and how acceptable and helpful the text program feels. A key focus is whether participants stay engaged, complete assessments, and find the intervention useful and safe, which are critical indicators of feasibility and acceptability for a future larger trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 24 *The age to provide consent in Nebraska is 19. Individuals recruited from the state of Nebraska must be 19 or older.
2. endorsement of past 2-week suicidal ideation
3. Resident of the United States
4. Owns a smartphone

Exclusion Criteria:

1. Serious mental illness for which intervention would be contraindicated (i.e., active psychosis or mania)
2. Imminent suicidality (i.e., experiencing active suicidal ideation with a plan and intent to act)
3. Written English language skills that are insufficient to engage in the consent, design, evaluation, or intervention procedures.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of suicidal thoughts | enrollment to 4 weeks
  The number of times an individual has experienced suicidal thoughts
Frequency of suicidal behaviors | enrollment to 4 weeks
  Frequency of suicidal behaviors
Severity of suicidal thoughts | enrollment to 4 weeks
  Severity of suicidal thoughts

SECONDARY OUTCOMES:
Unbearable Psychache Scale (UP3) | enrollment to 4 weeks
  Measure of psychic pain. Range 3-15. Higher scores indicate worse psychological pain.
Beck Hopelessness Scale-Short Form (BHS-SF) | Enrollment to 4 weeks
  Brief measure of hopelessness. Items rated 1 or 0. Scores range from 0-4, with higher scores indicating more hopelessness.
PROMIS Social Isolation - CAT | Enrollment to 4 weeks
  Brief measure of Social Isolation
Suicide Capacity Scale (SC3) | enrollment to 4 weeks
  Brief measure assessing subjective capacity to engage in suicide. Scores range from 0-36. Higher scores indicate greater suicide capacity
After-Scenario Questionnaire (ASQ) | enrollment to 4 weeks
  Brief measure assessing ease of use of the technology

OTHER OUTCOMES:
Suicide Related Coping Scale | Enrollment to 4 weeks
  Suicide Related Coping measure ranging from 0-68, higher scores indicate greater suicide related coping.

CONTACTS AND LOCATIONS:
Overall Officials: Jonah Meyerhoff, PhD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No